CLINICAL TRIAL: NCT02289664
Title: A Comparison of Coopdech, Intubrite, and CoPilot Video-laryngoscopes With Macintosh Laryngoscope for Tracheal Intubation in Pediatric Patients During Resuscitation. Randomized Crossover Manikin Trial
Brief Title: Videolaryngoscopy During Child Intubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Lukasz Szarpak, National Institute of Cardiology, Warsaw, Poland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ETI/2014/11
Record Dates: First submitted 2014-11-10; First posted 2014-11-13 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Cardiac Arrest
Keywords: intubation
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intubation without chest compressions (Experimental): Endotracheal intubation of pediatric mannikin during resuscitation without chest compressions.
  Interventions: Device: MAC; Device: Coopdech; Device: CoPilot; Device: Intubrite
- Intubation with uninterrupted chest compressions (Experimental): Endotracheal intubation of pediatric mannikin during resuscitation with uninterrupted chest compressions. In order to simulate the difficulties associated with intubation during uninterrupted chest compressions, CPR was performed by using LUCAS-2 (Physio-Control, Redmond, WA, U.S.).
  Interventions: Device: MAC; Device: Coopdech; Device: CoPilot; Device: Intubrite

INTERVENTIONS:
Device: MAC — Direct-Laryngoscopy
  Other Names: Macintosh Laryngoscope
Device: Coopdech — Video-Laryngoscopy -1
  Other Names: Coopdech Video Lartyngoscope Portable VLP-100
Device: CoPilot — Video-Laryngoscopy -2
  Other Names: CoPilot Video Laryngoscope
Device: Intubrite — Video-Laryngoscopy -3
  Other Names: Intubrite Video Laryngoscope System VLS 6600

SUMMARY:
We hypothesized that the video-laryngoscopes are beneficial for intubation of pediatric manikins while performing CPR. In the current study, we compared effectiveness of three video-laryngoscopes and Macintosh (MAC) laryngoscopes during pediatric resuscitation with and without chest compressions using an child manikin.

ELIGIBILITY:
Inclusion Criteria:

* Give voluntary consent to participate in the study
* minimum 1 year of work experience in health care

Exclusion Criteria:

* Not meet the above criteria
* Wrist or Low back diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-11; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Success of intubation | 1 MONTH
  effectiveness of first, second and third intubation attempts and overall effectiveness of intubation by participants using each device

SECONDARY OUTCOMES:
Intubation time | 1 MONTH
  time in seconds required for a successful intubation attempt
POGO score | 1 mONTH
  self-reported percentage of glottis opening (POGO) score
Cormack-Lehane grading | 1 MONTH
  self-reported percentage the vocal cord visualization using the Cormack-Lehane grading (grade 1-4)

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, Principal Investigator — Institute of Cardiology
Locations (1):
- International Institute of Rescue Research and Education, Warsaw, Masovia, Poland